CLINICAL TRIAL: NCT02918513
Title: WILD 5 Wellness: A 90-Day Intervention (WILD = Wellness Interventions for Life's Demands)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Saundra Jain, Adjunct Clinical Affiliate, School of Nursing, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-07-0021
Record Dates: First submitted 2016-07-25; First posted 2016-09-29 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Chronic Pain; Stress, Psychological; Healthy
Keywords: Wellness; Mental Wellness; Well-Being
MeSH Terms: conditions — Chronic Pain; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellness Intervention (Experimental): WILD 5 Wellness is an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition.
  Interventions: Behavioral: Wellness Element 1 - Exercise; Behavioral: Wellness Element 2 - Mindfulness; Behavioral: Wellness Element 3 - Sleep Hygiene; Behavioral: Wellness Element 4 - Social Connectedness; Behavioral: Wellness Element 5 - Nutrition; Behavioral: Wellness Element 6 - Wellness Exercises; Behavioral: Wellness Element 7 - Motivational Messages

INTERVENTIONS:
Behavioral: Wellness Element 1 - Exercise — 1. Daily wellness element focusing on Exercise; adherence documented online daily
Behavioral: Wellness Element 2 - Mindfulness — 2. Daily wellness element focusing on Mindfulness Meditation; adherence documented online daily
Behavioral: Wellness Element 3 - Sleep Hygiene — 3. Daily wellness element focusing on sleep hygiene; adherence documented online daily
Behavioral: Wellness Element 4 - Social Connectedness — 4. Daily wellness element focusing on Social Connectedness; adherence documented online daily
Behavioral: Wellness Element 5 - Nutrition — 5. Daily wellness element focusing on Nutrition; adherence documented online daily
Behavioral: Wellness Element 6 - Wellness Exercises — 6. Daily wellness workbook exercises focusing on improving mental wellness; adherence documented online daily
Behavioral: Wellness Element 7 - Motivational Messages — 7. Daily motivational emails offering information on one of the 5 wellness elements each day (Exercise, Mindfulness Meditation, Sleep, Social Connectedness, and Nutrition)

SUMMARY:
The purpose of this study is to explore the efficacy and feasibility of an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition.

DETAILED DESCRIPTION:
This study involves participating in a 90-day integrated, prescriptive, trackable wellness intervention, which includes five wellness elements: exercise, mindfulness, sleep, social connectedness, and nutrition.

The intervention is divided into three phases (each spanning 30-days): Phase 1 - 'Boot Camp', Phase 2 - Solidify, and Phase 3 - Sustain. Program requirements include: Implementing 5 wellness interventions daily for the first 30-days, at least 5 days for the next 30-days, and at least 3 days for the final 30-days, documenting daily online adherence, completing daily wellness exercises to improve mental wellness, and completing online program forms prior to beginning the program, at 30-days, and again at 90-days.

Once eligibility is confirmed via the initial orientation/screening call, study personnel will mail each participant a WILD 5 Wellness Workbook within one day of emailing participants their unique identification codes plus their start dates. Participants will be instructed to document adherence regarding their daily wellness practices and their daily wellness exercises online via Qualtrics, an online survey software. Participants can document their daily adherence using their computer and/or their smartphone as Qualtrics offers a mobile version of the Participant Tracking Form. A copy of the Participant Tracking Form will also be available in the WILD 5 Workbook so participants that prefer keeping a daily paper log can do so, and they can then transfer their program adherence information to the online Participant Tracking Form throughout the program. The workbook will contain the participant's personal identification code; no personal identification will appear in the workbook in order to protect participant confidentiality.

One day prior to a participant's start date, which will be set during the orientation/screening call, participants will receive an automated email from an online automated email service (MailChimp), with a reminder about their start date, and encouragement to contact study personnel with any questions or concerns.

Participants will also receive daily motivational emails from an online automated email service (MailChimp), which will provide general information about one of the five wellness elements and/or one of the wellness exercises, as well as encouragement to track their participation on a daily basis, and encouragement to contact study personnel via email with any questions and/or concerns.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older)
* English- speaking
* Access to a reliable Internet-enabled computer
* Possess basic computer skills
* Self-identify as having at least one of the health conditions listed on the online registration form or
* Self-identify as a community participant without a health condition.

Exclusion Criteria:

* Acutely suicidal and/or actively psychotic
* Non-English speaking
* Do not have access to an Internet-enabled computer
* Report a lack of basic computer skills
* Pregnant or plan to get pregnant during the next 90-days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | 0, 30, and 90 days - Primary endpoint is 30 days
  A self-reported depression scale used to assess severity of depression.
Change in Generalized Anxiety Disorder-7 (GAD-7) | 0, 30, and 90 days - Primary endpoint is 30 days
  A self-reported questionnaire used to assess anxiety symptoms.
Change in World Health Organization-5 (WHO-5) | 0, 30, and 90 days - Primary endpoint is 30 days
  A brief scale that measures mental well- being.
Change in The Mindful Attention Awareness Scale (MAAS) | 0, 30, and 90 days - Primary endpoint is 30 days
  A popular measure of mindfulness.
Change in The Sleep Condition Indicator (SCI) | 0, 30, and 90 days - Primary endpoint is 30 days
  A brief scale that evaluates insomnia disorder.
Change in The Social Connectedness Scale (SCS) | 0, 30, and 90 days - Primary endpoint is 30 days
  A brief scale that assesses the degree to which respondents feel connected to others.
Change in Eating and Appraisal Due to Emotions and Stress (EADES) | 0, 30, and 90 days - Primary endpoint is 30 days
  A scale assessing how individuals cope with and appraise stress in relation to food and eating.
Change in The Mediterranean-Dietary Approaches to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) | 0, 30, and 90 - Primary endpoint is 30 days
  A combination of the Mediterranean and DASH (Dietary Approaches to Stop Hypertension) diets shown to lower a person's risk of developing Alzheimer's disease.
Change in The Brief Pain Inventory (BPI) | 0, 30, and 90 days - Primary endpoint is 30 days
  A measurement tool for assessing clinical pain.
Change in The Sheehan Disability Scale (SDS) | 0, 30, and 90 days - Primary endpoint is 30 days
  A measurement tool for assessing functional impairment in three inter-related domains: work/school, social and family life.
Change in The Endicott Work Productivity Scale (EWPS) | 0, 30, and 90 days - Primary endpoint is 30 days
  A brief self-report questionnaire designed to obtain a sensitive measure of work productivity.
Change in Cognitive and Physical Functioning Questionnaire (CPFQ) | 0, 30, and 90 days - Primary endpoint is 30 days
  A brief scale that measures cognitive and executive dysfunction.
Change in The WILD 5 Wellness Scale (W5WS) | 0, 30, and 90 days - Primary endpoint is 30 days
  A brief scale designed specifically for this project to measure wellness.
Change in The WILD 5 Wellness Effort Scale (W5ES) | 0, 30, and 90 days - Primary endpoint is 30 days
  A scale designed specifically for this project to measure weekly adherence with program elements.
Change in The WILD 5 Wellness Elements Scale | 0, 30, and 90 days - Primary endpoint is 30 days
  A scale designed specifically for this project to measure elements of depression, anxiety, wellbeing, mindfulness, sleep quality, social connectedness, emotional eating, diet practices, pain, disability, work productivity, happiness, enthusiasm, resilience, and optimism.
The Post-Program Participant Questionnaire | 90 days
  A brief post study survey that captures participants' opinions about WILD 5 Wellness: 90-Day Intervention, and subjective ranking of their overall wellness.

CONTACTS AND LOCATIONS:
Overall Officials: Saundra M Jain, PsyD, LPC, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin School of Nursing, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cooney GM, Dwan K, Greig CA, Lawlor DA, Rimer J, Waugh FR, McMurdo M, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD004366. doi: 10.1002/14651858.CD004366.pub6. PMID 24026850
- [Result] Cruwys T, Dingle GA, Haslam C, Haslam SA, Jetten J, Morton TA. Social group memberships protect against future depression, alleviate depression symptoms and prevent depression relapse. Soc Sci Med. 2013 Dec;98:179-86. doi: 10.1016/j.socscimed.2013.09.013. Epub 2013 Sep 25. PMID 24331897
- [Result] Fardet A, Boirie Y. Associations between food and beverage groups and major diet-related chronic diseases: an exhaustive review of pooled/meta-analyses and systematic reviews. Nutr Rev. 2014 Dec;72(12):741-62. doi: 10.1111/nure.12153. Epub 2014 Nov 18. PMID 25406801
- [Result] Hui SK, Grandner MA. Associations between Poor Sleep Quality and Stages of Change of Multiple Health Behaviors among Participants of Employee Wellness Program. Prev Med Rep. 2015 Jan 1;2:292-299. doi: 10.1016/j.pmedr.2015.04.002. PMID 26046013
- [Result] Jeste DV, Palmer BW, Rettew DC, Boardman S. Positive psychiatry: its time has come. J Clin Psychiatry. 2015 Jun;76(6):675-83. doi: 10.4088/JCP.14nr09599. PMID 26132670
- [Result] Williams JM, Crane C, Barnhofer T, Brennan K, Duggan DS, Fennell MJ, Hackmann A, Krusche A, Muse K, Von Rohr IR, Shah D, Crane RS, Eames C, Jones M, Radford S, Silverton S, Sun Y, Weatherley-Jones E, Whitaker CJ, Russell D, Russell IT. Mindfulness-based cognitive therapy for preventing relapse in recurrent depression: a randomized dismantling trial. J Consult Clin Psychol. 2014 Apr;82(2):275-86. doi: 10.1037/a0035036. Epub 2013 Dec 2. PMID 24294837
- See also: Qualtrics security statement — https://www.qualtrics.com/security-statement/
- See also: Decision matrix: Cloud services — https://security.utexas.edu/iso-policies/cloud-services/decision-matrix
- See also: Online automated email service — http://www.mailchimp.com/
- See also: Program Overview Video — https://youtu.be/L_VIAnck05c